CLINICAL TRIAL: NCT04990193
Title: The Effect of Soft Orthoses and Strapping on Balance and Gait Performance in Children With Cerebral Palsy: A Randomized Controlled Trial
Brief Title: The Effect of Soft Orthoses on Balance and Gait Performance in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Ehab Mohamed Abd El Kafy, Professor of Physical Therapy, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-MED-1-0004
Record Dates: First submitted 2021-07-18; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Cerebral Palsy
Keywords: Balance; Gait; Strapping; Orthoses
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Children in the control group received the conventional physical therapy protocol which was designed to improve axial stability and trunk steadiness during standing and walking.
  Interventions: Other: Conventional Physical Therapy Protocol
- Study group (Experimental): The children in the study group received the conventional protocol given to the control group. Moreover, they wore TheraTog orthotic undergarment with its strapping system eight hours every day for twelve consecutive weeks.
  Interventions: Other: Conventional Physical Therapy Protocol; Other: TheraTog orthotic undergarment with its strapping system

INTERVENTIONS:
Other: Conventional Physical Therapy Protocol — The conventional physical therapy protocol was designed to improve axial stability and trunk steadiness during standing and walking. The conventional therapeutic protocol for every child was 3 sessions/week for 12 consecutive weeks. Every treatment session was conducted for 2 hours with a 15-minutes rest between the two training hours.
Other: TheraTog orthotic undergarment with its strapping system — TheraTog orthotic undergarment with its strapping system was applied for eight hours every day for twelve consecutive weeks.
  Arms: Study group

SUMMARY:
Most of the available studies that are relevant to motor rehabilitation for children with dyskinetic type of cerebral palsy are few and are comprised of small numbers of children. Further researches are necessary to explore new conservative therapeutic protocols and techniques that should contribute to control disorganized movement, handle postural asymmetry, maintain postural stability, and improve gait performance. Therefore, the objective of this study was to examine the effectiveness of soft orthosis and strapping system on balance, and gait performance in children with dyskinetic cerebral palsy.

DETAILED DESCRIPTION:
Dyskinetic type of cerebral palsy typically results from extrapyramidal and basal ganglia damage. The most common dyskinetic movement disorders are choreoathetosis and dystonia. Their clinical features include fluctuation of muscle tone, involuntary and in-coordinated movement, and posture instability. These features have significant negative impacts on the children's quality of life and performance of daily activities. Management strategy for children with dyskinesia requires both medical and rehabilitative treatment. Most of the available studies that are relevant to their motor rehabilitation are few and comprised of small numbers of children. The therapeutic modalities currently used for their rehabilitation require more evidence to certain their efficacy. Moreover, further researches are necessary to explore new conservative therapeutic protocols and techniques that should correct postural instability and improve the poor mobility of these children The objective of this study was to examine the effectiveness of an orthotic undergarment which is (TheraTog orthosis), and its strapping system on balance and gait performance in children with dyskinetic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Children of a confirmed diagnosis of dyskinetic cerebral palsy of choreoathetosis type were selected to participate in this study.
* Children (of both sexes) were between 12 and 16 years old were included .
* Their height and weight were more than 100 cm and 20 Kg respectively to be eligible for the evaluation process on the Biodex stability system.
* Children were able to comprehend and follow orders.
* Their gross motor development levels, as measured by Gross Motor Function Classification System, were between levels I and II.
* Throughout the study period, participating children were not subjected to any other physical therapy programs except the assigned treatment protocol.

Exclusion Criteria:

* Children were excluded from this study if they had inflexible spinal deformities interfering with spinal and limbs functional mobility.
* Children were also excluded if their skin were sensitive or inflamed to any materials used.
* Children who had seizures, perceptual disorders, visual problems, and auditory deficits did not participate as well.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change in the Overall Stability Indices {percentage value (%)} for Postural Stability Test (test that assessed the change in postural stability) | Data was collected at baseline, and 12 weeks after intervention commencement.
  The Biodex Balance System was used to assess the Change in the Overall Stability Indices of the Postural Stability Test. The test includes measurement of the following indices: overall stability index, anteroposterior index and mediolateral index which represents the children's ability to control their postural balance stability in all directions. High values % represent less stability and the children had difficulty in balance control. On the other hand lower values were indicative of a better balance control.
Change in the Pediatric Balance Scale score (scale that assessed the change in balance performance ) | Data was collected at baseline, and 12 weeks after intervention commencement.
  The Pediatric Balance Scale is a valid and reliable test to assess and re-assess balance deficits in children with mild and moderate motor disabilities. The test includes fourteen tasks that evaluate balance abilities and motor performance in children. 0-4 is the rating score for each item, where zero is the lowest score and 56 is the highest possible score for all tasks that indicate the best balance and motor performance ever.
Change in the gait parameter (step length) (This parameter indicated the change of gait performance). | Data was collected at baseline, and 12 weeks after intervention commencement.
  An electronic walkway that connected to a portable computer was used to measure the following gait parameter: step length (cm).
Change in the gait parameter (gait cycle time) (This parameter indicated the change of gait performance). | Data was collected at baseline, and 12 weeks after intervention commencement.
  An electronic walkway that connected to a portable computer was used to measure the following gait parameter: gait cycle time (seconds).
Change in the gait parameter (cadence) (This parameter indicated the change of gait performance). | Data was collected at baseline, and 12 weeks after intervention commencement.
  An electronic walkway that connected to a portable computer was used to measure the following gait parameter: cadence (steps/ minute).
Change in the gait parameter (velocity) (This parameter indicated the change of gait performance). | Data was collected at baseline, and 12 weeks after intervention commencement.
  An electronic walkway that connected to a portable computer was used to measure the following gait parameter: velocity (meter / second).

CONTACTS AND LOCATIONS:
Overall Officials: Ehab M Abd El Kafy, Ph.D, Principal Investigator — Faculty of Applied Medical Sciences - Umm Al Qura University
Locations (1):
- Umm Al Qura University, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No